CLINICAL TRIAL: NCT06293963
Title: Centering Equity in FDA Regulation: Front-of-package Food Label Effects in Latine and Limited English Proficiency Populations
Brief Title: Front-of-package Label Effects in Latine and Limited English Proficiency Populations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Duke University (Other); Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 24-0300a
Record Dates: First submitted 2024-02-27; First posted 2024-03-05 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2024-10

CONDITIONS: Diet, Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Numerical label (Experimental)
  Interventions: Behavioral: Guideline Daily Amounts label
- Interpretive text-only label (Experimental)
  Interventions: Behavioral: Interpretive text-only label
- Interpretive magnifying glass icon label (Experimental)
  Interventions: Behavioral: Interpretive magnifying glass icon label
- Separated interpretive magnifying glass icon label (Experimental)
  Interventions: Behavioral: Separated interpretive magnifying glass icon label

INTERVENTIONS:
Behavioral: Guideline Daily Amounts label — Labels that list the amount and percent of daily value of added sugar, sodium, or saturated fat, modeled after Guideline Daily Amounts labels.
  Arms: Numerical label
Behavioral: Interpretive text-only label — Interpretive text-only labels that state when a product contains high amounts of added sugar, sodium, or saturated fat.
  Arms: Interpretive text-only label
Behavioral: Interpretive magnifying glass icon label — Interpretive labels that state when a product contains high amounts of added sugar, sodium, or saturated fat, containing a magnifying glass icon.
  Arms: Interpretive magnifying glass icon label
Behavioral: Separated interpretive magnifying glass icon label — Interpretive labels that state when a product contains high amounts of added sugar, sodium, or saturated fat, containing a magnifying glass icon. Each nutrient will be on a separate label.
  Arms: Separated interpretive magnifying glass icon label

SUMMARY:
The goal of this experiment is to examine the effects of 4 types of front-of-package food labels among a sample of Latino adults. The main questions this experiment aims to answer are:

What front-of-package label design is most effective in helping Latino and low English proficiency consumers identify healthier and less healthy food products?

What front-of-package label design is most effective in helping Latino and low English proficiency consumers choose healthier food products?

Additionally, this experiment also aims to answer the following question:

Do the benefits of front-of-package label designs differ by English proficiency and parental status?

Participants will be randomly assigned to 1 of 4 types of front-of-package label designs and view their assigned label design on 3 sets of products. Each set will display 3 similar products, each high in either 1, 2, or 3 nutrients of concern. For each set, participants will select the product that they believe to be the healthiest, least healthy, and the product that they would most want to consume. Researchers will compare results across label designs.

DETAILED DESCRIPTION:
This study aims to determine which front-of-package label design is most effective at helping Latino consumers identify and choose healthier products, as well as explore whether the benefits of different front-of-package label designs differ by English proficiency. A Latino-focused panel company will recruit 4,000 US Latino adults of parental age (18-55 years), approximately 50% of whom will have limited English proficiency.

In a between-subjects experiment, researchers will randomize participants to 1 of 4 types of front-of-package label designs: a numerical label, an interpretive text-only label, an interpretive label with a magnifying glass icon, or separated interpretive labels with a magnifying glass icon. Participants will view their assigned label design on 3 similar products (each product high in either 1, 2, or 3 nutrients of concern) and complete selection tasks. These tasks will be repeated 3 times, each time with a different type of product (i.e., frozen meals, frozen pizzas, and frozen desserts), with the products displayed in random order.

ELIGIBILITY:
Inclusion Criteria:

* Identifying as Latino or Hispanic
* Ages 18-55 years old
* Residing in US

Exclusion Criteria:

* Not identifying as Latino or Hispanic
* Less than 18 or greater than 55 years old
* Not residing in the United States

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3306 (Actual)
Dates: Start 2024-08-09 (Actual); Primary Completion 2024-09-11 (Actual); Study Completion 2024-09-11 (Actual)

PRIMARY OUTCOMES:
Correct identification of healthiest product | During exposure to intervention (i.e., study stimuli), assessed during one-time online 10-minute survey.
  Correct identification of healthiest product will be measured by survey. Responses will be coded in a dichotomous 0-1 range, where 1 indicates that the participant correctly identified the healthiest product and 0 indicates that the participant incorrectly identified one of the other two less healthy products as the healthiest product.
Correct identification of least healthy product | During exposure to intervention (i.e., study stimuli), assessed during one-time online 10-minute survey.
  Correct identification of least healthy product will be measured by survey. Responses will be coded in a dichotomous 0-1 range, where 1 indicates that the participant correctly identified the least healthy product and 0 indicates that the participant incorrectly identified one of the other two healthier products as the least healthy product.

SECONDARY OUTCOMES:
Correct identification of products high in nutrients | During exposure to intervention (i.e., study stimuli), assessed during one-time online 10-minute survey.
  Correct identification of products high in nutrients (i.e., sugar, saturated fat, or sodium) will be measured by survey. Responses will be coded in a dichotomous 0-1 range, where 1 indicates that the participant correctly identified products that are high in a given nutrient and 0 indicates that the participant incorrectly identified products that are not high in a given nutrient as being high in such nutrient.
Selection of healthiest product for purchase | During exposure to intervention (i.e., study stimuli), assessed during one-time online 10-minute survey.
  Selection of healthiest product for purchase will be measured by survey. Responses will be coded in a dichotomous 0-1 range, where 1 indicates that the participant chose the healthiest product and 0 indicates that the participants selected one of the other two less healthy products.

CONTACTS AND LOCATIONS:
Overall Officials: Marissa G Hall, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- The University of North Carolina at Chapel Hill's Gillings School of Global Public Health, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
The Study Protocol and Statistical Analysis Plan will be shared prior to data collection. After data collection and analysis, a de-identified version of individual participant data and the analytic code will be shared through the Open Science Framework (OSF).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The Study Protocol and SAP will be available by mid-March 2024 (prior to data collection). IPD and analytic code will become available after data collection and analysis.
Access Criteria: Open access.

REFERENCES:
- [Derived] Hall MG, Lee CJY, Campos AD, Serrano N, Taillie LS, Falbe J, Musicus AA, Whitesell C, Martinez AV, Grummon AH. An RCT of Front-Of-Package Nutrition Labels in Latino Populations in the U.S. Am J Prev Med. 2025 Sep 20;70(3):108122. doi: 10.1016/j.amepre.2025.108122. Online ahead of print. PMID 40983259
- [Derived] Hall MG, Lee CJY, Campos AD, Serrano N, Taillie LS, Falbe J, Musicus A, Whitesell C, Martinez AV, Grummon AH. Effects of front-of-package nutrition labels in Latine and limited English proficiency populations: A randomized trial. medRxiv [Preprint]. 2025 May 11:2025.05.09.25327177. doi: 10.1101/2025.05.09.25327177. PMID 40385392

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-26): https://cdn.clinicaltrials.gov/large-docs/63/NCT06293963/Prot_SAP_002.pdf